CLINICAL TRIAL: NCT05115487
Title: Evaluation of Hand Functions in Newly Diagnosed Primary Sjögren's Syndrome Patients; A Controlled Cross-sectional Study
Brief Title: Evaluation of Hand Functions in Newly Diagnosed Primary Sjögren's Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Suleyman Akgol, M.D., Selcuk University
Other Study IDs: SJOGRENHAND
Record Dates: First submitted 2021-11-04; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Sjogren's Syndrome
MeSH Terms: conditions — Sjogren's Syndrome | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sjögren's syndrome: Subjects diagnosed with primary sjögren's syndrome according to the 2016 ACR/EULAR primary sjögren classification criteria will be included in the study.
  Interventions: Diagnostic Test: digital dynamometer
- Healthy controls
  Interventions: Diagnostic Test: digital dynamometer

INTERVENTIONS:
Diagnostic Test: digital dynamometer — Hand grip strength will be measured using a hand-held digital dynamometer with the patient sitting in a hard chair and elbow flexed to 90°. All assessments and measurements will be made by the same experienced physician blinded to patients' clinical data.
  Other Names: ultrasonography

SUMMARY:
Hand functions are decreased in rheumatic diseases such as systemic sclerosis and rheumatoid arthritis.

Sjögren's syndrome (SS) is a chronic systemic rheumatic disease characterized by lymphoplasmacytic infiltration of exocrine glands, especially salivary and lacrimal glands.

SS may be "primary" when it occurs alone (pSS) and "secondary" (sSS) when associated with another autoimmune disease. PSS is the most common connective tissue disease after rheumatoid arthritis and affects 0.3-3% of the population. Joint involvement is the most common involvement of pSS after sicca syndrome (50% of patients). Patients may have arthralgia with inflammatory features (morning stiffness > 30 minutes) or, less frequently, true symmetric polysynovitis mimicking rheumatoid arthritis (RA). The joint involvement of PSS is usually moderate (<5 affected joints) and mostly affects the small joints of the hands and upper extremities. PSS may also be responsible for myositis. Widespread pain, similar to primary fibromyalgia, is common in about 50 percent of patients with PSS.

The hand is one of the most important components affecting the functionality of the upper extremity. Grasping is one of the hand functions, for the continuity of daily living activities.

is an important function. Studies have shown that hand grip strength is correlated with upper extremity muscle strength, as well as general body muscle strength and pulmonary muscle strength.

As far as we know, hand functions have not been evaluated in newly diagnosed patients with pSS.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients aged 18-65 years diagnosed with Primary Sjogren's 2. Patients with normal cognitive functions

Exclusion Criteria:

* 1. Other connective tissue diseases other than primary Sjögren's 2.Pregnancy 3.Malignancy 4. Chronic diseases (DM, HT, Hypothyroidism, hyperthyroidism) 5. Cognitive disorder 6. Neurological or traumatic hand disorders leading to hand disorders (MS, Trauma, SVO) 7. Patients who have undergone major salivary gland surgery, have Graft Versus Host disease, have received Sarcoidosis, Head and Neck Radiotherapy, have a history of HTLV-1 or HIV

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed primary Sjögren's syndrome according to 2016 ACR/EULAR primary Sjögren classification criteria
Sampling Method: Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-12-07 (Estimated); Study Completion 2023-05-07 (Estimated)

PRIMARY OUTCOMES:
Hand grip strength | 1.5 years
  Hand grip strength will be measured by digital dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided